CLINICAL TRIAL: NCT03959163
Title: The Validity of the Quick Renal MRI in Pediatric Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-0492; A539800 (Other: UW Madison); SMPH/UROLOGY/UROLOGY (Other: UW Madison)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pyelonephritis; Pyelonephritis Acute; Renal Sclerosis
MeSH Terms: conditions — Pyelonephritis; Nephrosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- DMSA/Quick MRI (Other): All participants will go through DMSA and Quick MRI scan to help determine the validity of the Quick Renal MRI in pediatric kidney disease.
  Interventions: Diagnostic Test: Quick MRI

INTERVENTIONS:
Diagnostic Test: Quick MRI — A quick MRI scan takes about 15 mins or less. No IV or sedation will be necessary. The participant will be required to lie flat and still during the test. A parent will be allowed to be with the participant while they are in the scanner. The machine will produce loud intermittent sounds of banging or knocking so they will have to wear protective headphones. They can listen to music if they would like. If they are less than 1 year old, they will be swaddled and can be "held" during the test. If a child needs to have a parent in the scanner, it is ideal if the parent can have their head near the participant's legs and arms stretched out to hold the child's hands. If the parent needs to be by the patient's head, it can be accomplished by the parent lying head to head with the child or the parent lying on the child. Ideally they are lying head to head, or just outside of the scanner reaching in.

SUMMARY:
The investigators propose a new imaging method for children born with congenital anomalies of the urinary tract that is a rapid, injection-, sedation-, and radiation-free alternative: the quick renal MRI. This proposal hypothesizes that the quick renal MRI has high validity compared to current radiologic standard for renal infection and scarring, the 99mTechnetium-dimercaptosuccinic acid (99mTc- DMSA) renal scan in the detection of acute renal infections and scars. If the quick renal MRI is accurate, it could potentially replace the DMSA scan for those specific questions and ease the burden of testing for children with chronic renal disease. Findings from these studies will provide preliminary data and rationale for a multi-centered study to further test this new technology.

Participants will be 0-21 years of age and can expect to be on study for from 1 week (if enrolled in Aim 1) to 6 months (if enrolled in Aim 2).

DETAILED DESCRIPTION:
Children born with congenital anomalies of the urinary tract are susceptible to kidney infections and scarring. They form a high risk group for developing renal insufficiency in adulthood. A basic tenet in pediatric urology is that kidney infections should be prevented and otherwise promptly identified to minimize the risk of acquiring renal scars and permanent tissue damage.

The current radiologic standard for renal infection and scarring is the 99mTechnetium-dimercaptosuccinic acid (99mTc- DMSA) renal scan. This exam requires an intravenous injection, occurs over a 3 hour period, involves exposure to radiation, and can require sedation of young children. The investigators propose a new imaging method that is a rapid, injection-, sedation-, and radiation-free alternative: the quick renal MRI. This proposal hypothesizes that the quick renal MRI has high validity compared to the DMSA scan in the detection of acute renal infections and scars. If the quick renal MRI is accurate, it could potentially replace the DMSA scan for those specific questions and ease the burden of testing for children with chronic renal disease. Findings from these studies will provide preliminary data and rationale for a multi-centered study to further test this new technology.

There are two separate aims to this study, and study activities/schedule will vary depending on which aim the participant is in:

Aim 1: Inpatients presenting with acute pyelonephritis or possible acute pyelonephritis will be approached about the study. After participant's consent to the study, they will complete a clinical DMSA scan and quick MRI for the study. The DMSA scan and quick MRI will be completed within one week of each other, and ideally during the participant's inpatient stay.

Aim 2: Patients presenting to clinic for visits regarding their renal scarring will be approached about the study. If participant's consent to the study and if possible, they will schedule the quick MRI during this visit. The clinical DMSA scan and quick MRI should be completed within 6 months of each other for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1:

  * Patient is admitted to American Family Children's Hospital for a febrile UTI, suspected pyelonephritis, or diagnosed pyelonephritis
  * Undergoing clinical DMSA scan
* Aim 2:

  * Undergoing DMSA scans as a part of their routine clinical care
  * History of more than one UTI in the past year

Exclusion Criteria:

* Aim 1:

  * No evidence of pyuria on their urine analysis
  * Negative urine culture
  * Not comfortable with having a Quick MRI performed
* Both aims:

  * Contraindications to MRI

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Quick MRI as Compared to DMSA scan in Diagnosis of Suspected Acute Pyelonephritis | up to 1 week
  Children admitted for suspected acute pyelonephritis will undergo a clinical DMSA (gold-standard) renal scan and quick renal MRI to determine the sensitivity of this method.
  The sensitivity will be calculated with True Positive (TP) / TP + False Negative (FN)
Sensitivity of Quick MRI as compared to DMSA scan in Diagnosis of Renal Scars | up to 6 months
  To establish the sensitivity of the quick renal MRI compared to the DMSA scan (using DMSA as the 'gold standard') in the diagnosis of renal scars among children with recurrent UTI. Children with recurrent Urinary Tract Infection (UTI) will undergo a clinical DMSA renal scan and quick renal MRI. The sensitivity of the quick renal MRI to detect renal scars will be determined using DMSA as the standard.
  The sensitivity will be calculated with TP/TP+FN.
Specificity of Quick MRI as compared to DMSA scan in Diagnosis of Renal Scars | up to 6 months
  To establish the specificity of the quick renal MRI compared to the DMSA scan (using DMSA as the 'gold standard') in the diagnosis of renal scars among children with recurrent UTI. Children with recurrent UTI will undergo a clinical DMSA renal scan and quick renal MRI. The specificity of the quick renal MRI to detect renal scars will be determined using DMSA as the standard.
  The specificity will be calculated with True Negative (TN) / TN + False Positive (FP)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Cannon, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freedman AL; Urologic Diseases in America Project. Urologic diseases in North America Project: trends in resource utilization for urinary tract infections in children. J Urol. 2005 Mar;173(3):949-54. doi: 10.1097/01.ju.0000152092.03931.9a. PMID 15711347
- [Background] Hoberman A, Chao HP, Keller DM, Hickey R, Davis HW, Ellis D. Prevalence of urinary tract infection in febrile infants. J Pediatr. 1993 Jul;123(1):17-23. doi: 10.1016/s0022-3476(05)81531-8. PMID 8320616
- [Background] Sood A, Penna FJ, Eleswarapu S, Pucheril D, Weaver J, Abd-El-Barr AE, Wagner JC, Lakshmanan Y, Menon M, Trinh QD, Sammon JD, Elder JS. Incidence, admission rates, and economic burden of pediatric emergency department visits for urinary tract infection: data from the nationwide emergency department sample, 2006 to 2011. J Pediatr Urol. 2015 Oct;11(5):246.e1-8. doi: 10.1016/j.jpurol.2014.10.005. Epub 2015 Feb 7. PMID 26005017
- [Background] Copp HL, Halpern MS, Maldonado Y, Shortliffe LD. Trends in hospitalization for pediatric pyelonephritis: a population based study of California from 1985 to 2006. J Urol. 2011 Sep;186(3):1028-34. doi: 10.1016/j.juro.2011.04.101. Epub 2011 Jul 23. PMID 21784477
- [Background] Chen MJ, Cheng HL, Chiou YY. Risk factors for renal scarring and deterioration of renal function in primary vesico-ureteral reflux children: a long-term follow-up retrospective cohort study. PLoS One. 2013;8(2):e57954. doi: 10.1371/journal.pone.0057954. Epub 2013 Feb 28. PMID 23469116
- [Background] Rushton HG, Majd M. Dimercaptosuccinic acid renal scintigraphy for the evaluation of pyelonephritis and scarring: a review of experimental and clinical studies. J Urol. 1992 Nov;148(5 Pt 2):1726-32. doi: 10.1016/s0022-5347(17)37014-3. PMID 1331545
- [Background] Hari P, Bagga A. Antimicrobial prophylaxis for children with vesicoureteral reflux. N Engl J Med. 2014 Sep 11;371(11):1071-2. doi: 10.1056/NEJMc1408559. No abstract available. PMID 25207775
- [Background] Faust WC, Diaz M, Pohl HG. Incidence of post-pyelonephritic renal scarring: a meta-analysis of the dimercapto-succinic acid literature. J Urol. 2009 Jan;181(1):290-7; discussion 297-8. doi: 10.1016/j.juro.2008.09.039. Epub 2008 Nov 14. PMID 19013606
- [Background] Rushton HG, Majd M, Jantausch B, Wiedermann BL, Belman AB. Renal scarring following reflux and nonreflux pyelonephritis in children: evaluation with 99mtechnetium-dimercaptosuccinic acid scintigraphy. J Urol. 1992 May;147(5):1327-32. doi: 10.1016/s0022-5347(17)37555-9. PMID 1314912
- [Background] Lee LC, Lorenzo AJ, Koyle MA. The role of voiding cystourethrography in the investigation of children with urinary tract infections. Can Urol Assoc J. 2016 May-Jun;10(5-6):210-214. doi: 10.5489/cuaj.3610. PMID 27713802
- [Background] Fillion ML, Watt CL, Gupta IR. Vesicoureteric reflux and reflux nephropathy: from mouse models to childhood disease. Pediatr Nephrol. 2014 Apr;29(4):757-66. doi: 10.1007/s00467-014-2761-3. Epub 2014 Feb 6. PMID 24500705
- [Background] McKibben MJ, Seed P, Ross SS, Borawski KM. Urinary Tract Infection and Neurogenic Bladder. Urol Clin North Am. 2015 Nov;42(4):527-36. doi: 10.1016/j.ucl.2015.05.006. Epub 2015 Jul 7. PMID 26475949
- [Background] Oakeshott P, Hunt GM, Poulton A, Reid F. Expectation of life and unexpected death in open spina bifida: a 40-year complete, non-selective, longitudinal cohort study. Dev Med Child Neurol. 2010 Aug;52(8):749-53. doi: 10.1111/j.1469-8749.2009.03543.x. Epub 2009 Dec 9. PMID 20015251
- [Background] Woodhouse CR. Myelomeningocele in young adults. BJU Int. 2005 Feb;95(2):223-30. doi: 10.1111/j.1464-410X.2005.05374.x. No abstract available. PMID 15667645
- [Background] Wang HH, Lloyd JC, Wiener JS, Routh JC. Nationwide Trends and Variations in Urological Surgical Interventions and Renal Outcome in Patients with Spina Bifida. J Urol. 2016 Apr;195(4 Pt 2):1189-94. doi: 10.1016/j.juro.2015.11.033. Epub 2016 Feb 28. PMID 26926542
- [Background] Ouyang L, Bolen J, Valdez R, Joseph D, Baum MA, Thibadeau J. Characteristics and survival of patients with end stage renal disease and spina bifida in the United States renal data system. J Urol. 2015 Feb;193(2):558-64. doi: 10.1016/j.juro.2014.08.092. Epub 2014 Aug 25. PMID 25167993
- [Background] Routh JC, Cheng EY, Austin JC, Baum MA, Gargollo PC, Grady RW, Herron AR, Kim SS, King SJ, Koh CJ, Paramsothy P, Raman L, Schechter MS, Smith KA, Tanaka ST, Thibadeau JK, Walker WO, Wallis MC, Wiener JS, Joseph DB. Design and Methodological Considerations of the Centers for Disease Control and Prevention Urologic and Renal Protocol for the Newborn and Young Child with Spina Bifida. J Urol. 2016 Dec;196(6):1728-1734. doi: 10.1016/j.juro.2016.07.081. Epub 2016 Jul 27. PMID 27475969
- [Background] MacKenzie JR. A review of renal scarring in children. Nucl Med Commun. 1996 Mar;17(3):176-90. doi: 10.1097/00006231-199603000-00002. PMID 8692483
- [Background] Michaud JE, Gupta N, Baumgartner TS, Kim B, Bosemani T, Wang MH. Cost and radiation exposure in the workup of febrile pediatric urinary tract infections. J Surg Res. 2016 Jun 15;203(2):313-8. doi: 10.1016/j.jss.2016.03.042. Epub 2016 Mar 26. PMID 27363638
- [Background] Iskandar BJ, Sansone JM, Medow J, Rowley HA. The use of quick-brain magnetic resonance imaging in the evaluation of shunt-treated hydrocephalus. J Neurosurg. 2004 Nov;101(2 Suppl):147-51. doi: 10.3171/ped.2004.101.2.0147. PMID 15835101
- [Background] Rozovsky K, Ventureyra EC, Miller E. Fast-brain MRI in children is quick, without sedation, and radiation-free, but beware of limitations. J Clin Neurosci. 2013 Mar;20(3):400-5. doi: 10.1016/j.jocn.2012.02.048. Epub 2012 Dec 21. PMID 23266077
- [Background] Yue EL, Meckler GD, Fleischman RJ, Selden NR, Bardo DM, Chu O'Connor AK, Vu ET, Fu R, Spiro DM. Test characteristics of quick brain MRI for shunt evaluation in children: an alternative modality to avoid radiation. J Neurosurg Pediatr. 2015 Apr;15(4):420-6. doi: 10.3171/2014.9.PEDS14207. Epub 2015 Jan 30. PMID 25634816
- [Background] Christy A, Murchison C, Wilson JL. Quick Brain Magnetic Resonance Imaging With Diffusion-Weighted Imaging as a First Imaging Modality in Pediatric Stroke. Pediatr Neurol. 2018 Jan;78:55-60. doi: 10.1016/j.pediatrneurol.2017.09.020. Epub 2017 Oct 9. PMID 29174005
- [Background] Sheridan DC, Newgard CD, Selden NR, Jafri MA, Hansen ML. QuickBrain MRI for the detection of acute pediatric traumatic brain injury. J Neurosurg Pediatr. 2017 Feb;19(2):259-264. doi: 10.3171/2016.7.PEDS16204. Epub 2016 Nov 25. PMID 27885947
- [Background] Thompson EM, Baird LC, Selden NR. Results of a North American survey of rapid-sequence MRI utilization to evaluate cerebral ventricles in children. J Neurosurg Pediatr. 2014 Jun;13(6):636-40. doi: 10.3171/2014.2.PEDS13567. Epub 2014 Apr 11. PMID 24724716
- [Background] Kovanlikaya A, Okkay N, Cakmakci H, Ozdogan O, Degirmenci B, Kavukcu S. Comparison of MRI and renal cortical scintigraphy findings in childhood acute pyelonephritis: preliminary experience. Eur J Radiol. 2004 Jan;49(1):76-80. doi: 10.1016/S0720-048X(02)00350-9. PMID 14975495
- [Background] Weller A, Barber JL, Olsen OE. Gadolinium and nephrogenic systemic fibrosis: an update. Pediatr Nephrol. 2014 Oct;29(10):1927-37. doi: 10.1007/s00467-013-2636-z. Epub 2013 Oct 22. PMID 24146299
- [Background] Aoyagi J, Odaka J, Kuroiwa Y, Nakashima N, Ito T, Saito T, Kanai T, Yamagata T, Momoi MY. Utility of non-enhanced magnetic resonance imaging to detect acute pyelonephritis. Pediatr Int. 2014 Jun;56(3):e4-6. doi: 10.1111/ped.12312. PMID 24894941
- [Background] Verswijvel G, Vandecaveye V, Gelin G, Vandevenne J, Grieten M, Horvath M, Oyen R, Palmers Y. Diffusion-weighted MR imaging in the evaluation of renal infection: preliminary results. JBR-BTR. 2002 Apr-May;85(2):100-3. PMID 12083620
- [Background] Rathod SB, Kumbhar SS, Nanivadekar A, Aman K. Role of diffusion-weighted MRI in acute pyelonephritis: a prospective study. Acta Radiol. 2015 Feb;56(2):244-9. doi: 10.1177/0284185114520862. Epub 2014 Jan 17. PMID 24443116
- [Background] De Pascale A, Piccoli GB, Priola SM, Rognone D, Consiglio V, Garetto I, Rizzo L, Veltri A. Diffusion-weighted magnetic resonance imaging: new perspectives in the diagnostic pathway of non-complicated acute pyelonephritis. Eur Radiol. 2013 Nov;23(11):3077-86. doi: 10.1007/s00330-013-2906-y. Epub 2013 Jun 8. PMID 23749224
- [Background] Vivier PH, Sallem A, Beurdeley M, Lim RP, Leroux J, Caudron J, Coudray C, Liard A, Michelet I, Dacher JN. MRI and suspected acute pyelonephritis in children: comparison of diffusion-weighted imaging with gadolinium-enhanced T1-weighted imaging. Eur Radiol. 2014 Jan;24(1):19-25. doi: 10.1007/s00330-013-2971-2. Epub 2013 Jul 25. PMID 23884301
- [Background] Chan YL, Chan KW, Yeung CK, Roebuck DJ, Chu WC, Lee KH, Metreweli C. Potential utility of MRI in the evaluation of children at risk of renal scarring. Pediatr Radiol. 1999 Nov;29(11):856-62. doi: 10.1007/s002470050713. PMID 10552069
- [Background] Kavanagh EC, Ryan S, Awan A, McCourbrey S, O'Connor R, Donoghue V. Can MRI replace DMSA in the detection of renal parenchymal defects in children with urinary tract infections? Pediatr Radiol. 2005 Mar;35(3):275-81. doi: 10.1007/s00247-004-1335-0. Epub 2004 Oct 14. PMID 15490148